CLINICAL TRIAL: NCT00102622
Title: Phase I of Phase I/II Randomized Study of Intraperitoneal tgDCC-E1 and Intravenous Paclitaxel in Women With Platinum-Resistant Ovarian Cancer
Brief Title: Intraperitoneal tgDCC-E1 and Intravenous Paclitaxel in Women With Platinum-Resistant Ovarian Cancer
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Phase I/II study that did not progress to Phase II
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ID02-321; P50CA083639 (NIH); NCT02157870 (obsolete NCT alias)
Record Dates: First submitted 2005-01-31; First posted 2005-02-01 (Estimated); Last update posted 2018-11-13 (Actual); Status verified 2018-11

CONDITIONS: Ovarian Cancer
Keywords: Ovary; ovarian cancer; biologic therapy; platinum-resistant; platinum-refractory ovarian cancer; platinum-resistant ovarian cancer; paclitaxel; tgDCC-E1A; E1A; Taxol
MeSH Terms: conditions — Ovarian Neoplasms | interventions — Paclitaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm 1: Paclitaxel + tgDCC-E1A (Experimental): 80 mg/m^2 intravenous Paclitaxel and intraperitoneal (IP) tgDCC-E1A starting dose 1.8 mg DNA/m^2 weekly for six treatments every 7 days.
  Interventions: Biological: Intraperitoneal tgDCC-E1A; Drug: Paclitaxel
- Arm 2: Paclitaxel Alone (Active Comparator): Weekly single agent intravenous Paclitaxel 80 mg/m^2 for six treatments every 7 days.
  Interventions: Drug: Paclitaxel

INTERVENTIONS:
Biological: Intraperitoneal tgDCC-E1A — Starting Dose Level: 1.8 mg DNA/m^2 intraperitoneal every 7 days +/- 2 days for a total of 6 treatments each cycle.
  Other Names: E1A
  Arms: Arm 1: Paclitaxel + tgDCC-E1A
Drug: Paclitaxel — 80 mg/m^2 intravenous (IV) every 7 days +/- 2 days for a total of 6 treatments.
  Other Names: Taxol

SUMMARY:
The goal of this clinical research study is to find the highest safe dose of intraperitoneal tgDCC-E1A that can be given in combination with paclitaxel as a treatment for patients with recurrent, platinum-resistant ovarian cancer. How the cancer responds to this treatment will also be studied. Researchers will also ask the patients if they will allow additional tumor samples to be collected and extra blood samples to be drawn. These samples will be used to learn about the biological response before and after treatment.

DETAILED DESCRIPTION:
Primary Objective

* To evaluate toxicity and establish the maximum tolerated dose (MTD) of intraperitoneal tgDCC-E1A in combination with intravenous paclitaxel.
* To measure tumor response of intraperitoneal tgDCC-E1A in combination with intravenous paclitaxel and compare to intravenous paclitaxel

Secondary Objective

* To measure time to progression and overall survival.
* To examine the biological effects of combined tgDCC- E1A and paclitaxel in ovarian cancer cells as measured by laboratory testing.

Epithelial ovarian cancer is a significant public health problem. It is the sixth most common cancer in women worldwide. Globally, it is estimated that 162,000 new cases are diagnosed per year, and that 106,000 women die from the disease per year.

Signs and symptoms of ovarian cancer are often subtle. Seventy-five percent of subjects will present with advanced stage III and IV disease. Standard treatment for stage III/IV subjects consists of surgical debulking to the maximal extent possible and chemotherapy with paclitaxel plus a platinum compound (cisplatin or carboplatin). Despite high initial response rates, the overall survival for this group is poor, with only 20% of stage III and less than 5% of stage IV subjects surviving five years.

Treatment of recurrent ovarian cancer varies depending upon the interval between prior treatment and recurrence. Twenty percent of subjects are classified as "platinum-refractory", in that they fail to have even a partial response to a platinum-containing regimen. Subjects with recurrent or progressive disease less than six months after initial therapy have a poor response rate to repeat treatment with a platinum-containing regimen, and are generally considered to have "platinum-resistant" disease. In contrast, subjects with recurrent disease greater than six months after initial therapy have better response rates to repeat treatment with platinum-containing regimens, and are generally considered to have "platinum-sensitive" disease.

There is no consensus for the treatment of "platinum-refractory" or "platinum-resistant" ovarian cancer, a class of individuals who are particularly challenging to treat. Prognosis is poor, and treatment is primarily palliative in nature. Responses to a variety of single chemotherapeutic agents, as well as to a combination of agents in largely phase II trials have been similar, ranging from 10-35%. Intravenous (IV) paclitaxel, given alone or in combination with other agents is a standard treatment for subjects who have relapsed. In an attempt to increase the dose intensity of paclitaxel therapy, weekly IV paclitaxel has been recommended. This treatment schedule is well tolerated, but the response rate in heavily pretreated subjects is still only 28.9%.

Given that this group of subjects is poorly responsive to conventional chemotherapy, and consequently has limited options, an alternative approach to treatment is warranted. The use of a gene therapy agent with anti-tumor effects and the ability to sensitize cancer cells to traditional chemotherapy is appealing.

* Overview of the Effect of E1A Gene Transfer on Cancer Cells:

E1A, a gene derived from Adenovirus type 5, has been shown to have potent anti-neoplastic activity through a variety of mechanisms, including down-regulation of HER-2/neu overexpression, induction of apoptosis, inhibition of metastasis, and reversion of tumor cells toward a differentiated epithelial phenotype. The E1A gene has also been shown to have an additive effect in vitro and in vivo on the apoptosis induced by chemotherapy and radiotherapy. The E1A gene has been successfully transfected into human cells both in vitro and in vivo using tgDCC-E1A (E1A-Lipid Complex), which consists of the E1A plasmid (pE1A-K2) complexed to the cationic lipid gene delivery system comprised of DC-Cholesterol 3b[N-(N'N'-dimethylaminoethane)-carbamoyl] cholesterol hydrochloride and DOPE (1,2-dioleoyl-sn-glycero-3-phosphoethanolamine).

* Rationale for Use of Cationic Lipids to Deliver DNA:

Cationic lipids can form complexes with negatively charged DNA plasmids and facilitate the transfer of genes to target cells. They are useful agents for delivery of gene therapy because they are synthesized chemically, are simple to manufacture, and pose no infectious risk. The cationic derivative of cholesterol, 3b[N-(N'N'-dimethylaminoethane)-carbamoyl] cholesterol hydrochloride (DC-Chol) is an ideal cationic lipid for therapeutic use, as the cationic charge is provided by a non-toxic tertiary amine with a biodegradable carbamoyl bond. DC-Chol can be used to prepare liposomes in combination with the neutral 1,2-dioleoyl-sn-glycero-3-phosphoethanolamine (DOPE) with a DC-Chol to DOPE ratio of 6:4. This liposome combination can be mixed with a plasmid encoding E1A to form tgDCC-E1A.

The final preparation of tgDCC-E1A can be made within a range of lipid:DNA ratios, all of which have been shown in cell culture and in animal models to result in expression of E1A. Clinical trials of tgDCC-E1A for injection into solid tumors have used a final preparation with a lipid:DNA ratio of 1 nmol lipid to 1 microgram DNA [tgDCC-E1A (1:1)]. Early clinical trials evaluating intracavitary administration (e.g. intraperitoneal infusion for ovarian cancer) used a preparation with a lipid:DNA ratio of 10 nmol lipid to 1 microgram DNA [tgDCC-E1A (10:1)]. More recent protocols of intraperitoneal delivery for ovarian cancer have used a preparation with a lipid:DNA ratio of 3 nmol lipid to 1 microgram DNA [tgDCC-E1A (3:1)], as will this protocol.

* Rationale for Intraperitoneal Delivery of tgDCC-E1A:

The peritoneal cavity is a common site of tumor recurrence after initial "radical" surgical treatment of ovarian malignancies. Dissemination in this cavity is often widespread. Because of the unusual natural course of ovarian cancer (characterized by its tendency to be confined to the peritoneal cavity), control of metastatic disease in the peritoneal cavity is an important and challenging problem, which can be improved by direct delivery of drug into the peritoneal cavity.

ELIGIBILITY:
Inclusion Criteria:

* Age greater than or equal to 18 years
* Recurrent epithelial ovarian cancer or primary peritoneal cancer with histologic confirmation of the original tumor. Recurrent disease may be manifested as an elevated cancer antigen (CA)-125 using the following criteria: (a) increase in CA-125 to at least 2 times the upper limit of normal (assayed on 2 occasions at least 7 days apart) for subjects with a history of normal pre-treatment values or values that normalized with the most recent treatment - OR - (b) increase in CA-125 to 2 times the lowest observed value on the most recent treatment (assayed on two occasions at least 7 days apart) for subjects whose CA-125 did not normalize with the most recent treatment.
* Platinum-resistant disease, defined as recurrence less than six months after discontinuation of treatment with platinum therapy or platinum-refractory disease defined as progression on a platinum-containing regimen.
* A treatment-free interval of at least three weeks for cytotoxic therapies, radiation therapy, or other experimental drugs prior to first treatment on this protocol.
* A Zubrod performance status of two or less.

Exclusion Criteria:

* Previous administration of tgDCC-E1A.
* Progression on any taxane-containing regimen, or recurrent within 6 months of receiving a weekly taxane-containing regimen.

Previous radiation to more than 25% of marrow-bearing areas.

* Any of the following laboratory values: Hemoglobin <9.0 gm/dl, absolute neutrophil count (ANC) <1.5 K/ml, platelet <100 K/ml, creatinine >2 mg/dl, bilirubin >2 mg/dl, Aspartate Aminotransferase (AST) or Alanine Aminotransferase (ALT)>2 times the upper limit of normal, or abnormal coagulation profiles (>2 seconds beyond upper range of normal Prothrombin Time (PT) or Partial thromboplastin time (PTT)).
* Known human immunodeficiency virus (HIV)-positive status or active systemic infection.
* History of other invasive malignancies, except for non-melanoma skin cancer, unless there is no evidence of other cancer within the past 5 years.
* Patients with grade 2 or greater neurotoxicity.
* Patients with unstable angina or those who have had a myocardial infarction within the past six months. Patients with evidence of abnormal cardiac conduction are eligible if their disease has been stable for the past six months. Patients with an ejection fraction under 40%.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2004-12-01 (Actual); Primary Completion 2012-07 (Actual); Study Completion 2012-07 (Actual)

PRIMARY OUTCOMES:
Maximum Tolerated Dose (MTD) of Intraperitoneal (IP) tgDCC-E1A in combination with Intravenous (IV) Paclitaxel | 6 week cycle (cycle consists of 6 weekly treatments)
  Dose combinations assigned using the Continuous Reassessment Method (CRM) with up to 8 cohorts of three subjects each assigned to one of the three tgDCC-E1A dose combinations (1.8 , 3.6 or 5.0 mg DNA/m^2). Three weeks after third subject started treatment, the number of subjects who experienced dose limiting toxicities (DLT) tabulated. The next cohort of three subjects assigned to same or next higher dose combination using a computer algorithm that evaluates proportion of subjects who experienced a DLT.

SECONDARY OUTCOMES:
Tumor response of intraperitoneal (IP) tgDCC-E1A in combination with intravenous (IV) paclitaxel compared to IV paclitaxel alone | 5 Years
  Response Evaluation Criteria in Solid Tumors (RECIST): Complete Response: disappearance all target & non-target lesions, no evidence new lesions in 2 disease assessments 4 weeks apart; Partial Response (PR): >30% decrease in sum longest dimensions (LD) of all target measurable lesions reference baseline sum of LD; 2 disease assessments 4 weeks apart required. IF ONLY target lesion is solitary pelvic mass measured by physical exam, not radiographically measurable, 50% decrease in LD required; Progressive disease (PD): >20% increase in sum LD of target lesions references smallest sum LD or appearance new lesions. IF ONLY target lesion is solitary pelvic mass measured by physical exam, not radiographically measurable, 50% increase in LD required; Stable disease: neither sufficient shrinkage for PR nor increase for PD, reference smallest sum LD since treatment started, or IF non-target lesions persistence of 1+ non-target lesions and/or maintenance of tumor marker above normal limits.

CONTACTS AND LOCATIONS:
Overall Officials: Naoto Ueno, MD, PHD, Principal Investigator — UT MD Anderson Cancer Center
Locations (1):
- University of Texas M. D. Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: The University of Texas MD Anderson Cancer Center official website — http://www.mdanderson.org